CLINICAL TRIAL: NCT00421616
Title: A Diet Higher in Animal-Based Protein is More Effective in Promoting Weight Loss in Overweight and Obese Individuals Than Other Protein Based Diets.
Brief Title: Effectiveness of High Protein Diets in Promoting Weight Loss in Overweight and Obese Subjects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Wollongong (Other)
Collaborators: National Centre of Excellence in Functional Foods, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE06/332
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Overweight
Keywords: Calorimetry; Overweight; Weight loss; Appetite
MeSH Terms: conditions — Overweight; Weight Loss

INTERVENTIONS:
Behavioral: High protein diet study

SUMMARY:
Several studies have reported greater weight loss when following high meat-protein diets but limited studies have studied high plant-based protein diets. Thus we aim to investigate the effect of high protein diets in weight management and also to investigate the superior protein source in achieving this effect. In addition, we aim to develop dietary intervention strategies that are realistic and sustainable.

DETAILED DESCRIPTION:
Participants will be randomised to either high-protein diets (30% of energy) from animal or plant sources or standard protein diet (15% of energy) weight loss diet for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese
* Age 18 and above
* Both males and females
* Live in Illawarra Area of Australia

Exclusion Criteria:

* Regular medication
* Smoker
* Food allergies
* Presence of disease which may alter metabolic rate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2007-02

PRIMARY OUTCOMES:
Weight & anthropometric measurements at 0 and 3 months
Energy expenditure
Substrate oxidation
Compliance to diets

SECONDARY OUTCOMES:
Blood lipids
Appetite

CONTACTS AND LOCATIONS:
Overall Officials: Marijka Batterham, PhD, Principal Investigator — Smart Foods Centre, University of Wollongong; Linda Tapsell, PhD, Principal Investigator — National Centre of Excellence in Functional Foods, Australia; Arthur Jenkins, PhD, Principal Investigator — School of Health Sciences, University of Wollongong
Locations (1):
- Smart Foods Centre, University of Wollongong, Wollongong, New South Wales, Australia

REFERENCES:
- [Derived] Tan SY, Batterham M, Tapsell L. Activity counts from accelerometers do not add value to energy expenditure predictions in sedentary overweight individuals during weight loss interventions. J Phys Act Health. 2011 Jul;8(5):675-81. doi: 10.1123/jpah.8.5.675. PMID 21734313